CLINICAL TRIAL: NCT05568823
Title: Biomarkers of ANTidepressant RESponse and Development Risk of Bipolar Disorder
Acronym: ANTaRES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-51
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Depression, Bipolar; Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Stratification on two groups of patients subsequently identified as responders or non-responders, after 8 weeks of treatment. Patients will be classified as responders or non-responders on the basis of the evolution of the MADRS depression scale score, i.e. an improvement of more than 50% in the intensity of symptoms between the beginning of the treatments and 8 weeks afterwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients "responding" to treatment after 8 weeks of treatment (Other): Patients "responding" to treatment after 8 weeks of treatment: i.e. whose clinical evolution is beneficial.
  Interventions: Other: Blood sampling
- Patients "non-responding" to treatment after 8 weeks of treatment (Other): Patients "non-responding" to treatment after 8 weeks of treatment: i.e. whose clinical evolution is not satisfactory.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Measurement of markers of disease evolution
  Other Names: Psychiatric survey; MRI Exam

SUMMARY:
One in five people will present a major depressive episode (MDE) in their lifetime. While antidepressants (ADs) are currently the standard treatment for MDE, the first AD prescribed is effective in less than 40% of patients and a complete clinical response is only observed after several weeks. Identifying early biomarkers of the response to treatment with an AD could allow the clinician to rapidly identify patients in whom treatment will not be effective and therefore modify patient care. We have recently shown that the messenger RNA (mRNA) of two proteins, ELK1 and GPR56, were present in different amounts in the blood cells of "responder" compared to those of "non-respondent" patients. In this context, our main objective will be to determine whether ELK1 and GPR56 mRNAs, are very early biomarkers of the response to AD, i.e., biomarkers whose variation precedes the clinical response by several weeks. Secondary objectives will be to identify early phase changes in neurophysiological measures, cognitive and behavioral tasks, as well as levels of blood coding and non-coding RNAs, serum cytokine, mitochondrial and metabolic markers, neuroimaging markers as biomarkers of differential treatment outcomes to antidepressant treatment.

Patients will be treated with SERTRALINE or FLUOXETINE or DULOXETINE or MAPROTILINE (in monotherapy) with or without adjunct benzodiazepine.

Patients are identified as responders or non-responders based on their clinical assessment at 8 weeks after treatment onset.

In addition, a second stage will collect data to address another important issue for the management of patients with a MDE: to discriminate those with a major depressive disorder (MDD) from those with a bipolar disorder (BD). BD diagnosis is one of the most common reasons of failure to response to ADs. Therefore, one of our secondary objectives will be to identify biomarkers to differentiate between these two categories of patients. To do this, we will follow patients for a period of 24 months to identify those who will present during this follow-up the diagnostic criteria of bipolarity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient between 18 and 65 years of age
* Sufficient knowledge of the French language to complete the assessments
* Inpatients or outpatients with a major depressive episode (DSM-5 criteria);
* Score above 19 on the MADRS depression scale (moderate to severe depression);
* Without antidepressants, mood stabilizers or antipsychotics treatment or having stopped the previous medication(s) for more than 5 times the half-life of the prescribed treatment(s);
* Eligible for antidepressant monotherapy with SERTRALINE or FLUOXETINE or DULOXETINE or MAPROTILINE, with or without benzodiazepine therapy, and in whom treatment is feasible within days of inclusion.

Exclusion Criteria:

* • Patient with bipolar disorder, schizophrenia or psychotic disorder as defined by the DSM-5 and assessed by the MINI or any other pathology or treatment deemed clinically incompatible with the study by the investigator;

  * Patient with moderate to severe substance use disorders (>=4/11 criteria as defined in the DSM-5) and with the exception of smoking disorders
  * Patient with pregnancy, unstable physiological condition or severe and symptomatic medical condition;
  * Patient with a diagnosed neurological disorder affecting central nervous system function;
  * Patient unable to give informed consent to participate in this study or unable to give the volunteer informed information;
  * Patient who are not covered by a social security system;
  * Patient under court protection or guardianship
  * Patient who have received a vaccination within one month prior to initiation of treatment or who plan to be vaccinated within 2 weeks of initiation of treatment > For patient undergoing MRI: presence of a contraindication for MRI examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
Predictive value for antidepressant response of ELK1 mRNA levels or changes 3 days after AD start | 8 weeks of treatment
  The area under the curve (AUC) value determined by receiving operating characteristic (ROC) analysis of ELK1 mRNA levels for the evolution of psychiatric symptoms following AD start, during a 8-weeks follow-up. Patients are identified as responders or nonresponders based on their clinical assessment

SECONDARY OUTCOMES:
Predictive value for antidepressant response of GPR56 and ELK1 mRNA levels at baseline, 3 days, 2 weeks or 8 weeks after AD start | 8 weeks of treatment
  The area under the curve (AUC) value determined by receiving operating characteristic (ROC) analysis of GPR56 and ELK1 ELISA tests from whole blood for the evolution of psychiatric symptoms following AD start, during a 8-weeks follow-up. Patients are identified as responders or nonresponders based on their clinical assessment
Predictive value for antidepressant response of coding and non-coding (micro, circular, long non coding) RNA blood levels at baseline, 3 days, 2 weeks or 8 weeks after AD start | 8 weeks of treatment
  The area under the curve (AUC) value determined by receiving operating characteristic (ROC) analysis of coding and non-coding (micro, circular, long non coding) blood RNA levels for the evolution of psychiatric symptoms following AD start, during a 8-weeks follow-up. Patients are identified as responders or nonresponders based on their clinical assessment
Predictive value for antidepressant response of serum cytokine concentration measured by immunoassay at baseline, 3 days, 2 weeks or 8 weeks, after AD start | 8 weeks of treatment
  The area under the curve (AUC) value determined by receiving operating characteristic (ROC) analysis of serum cytokine concentration measured by immunoassay for the evolution of psychiatric symptoms following AD start, during a 8-weeks follow-up. Patients are identified as responders or nonresponders based on their clinical assessment
Predictive value for antidepressant response of peripheral mitochondrial markers at baseline, 3 days 2 weeks or 8 weeks, after AD start Time Frame: 8 weeks of treatment | 8 weeks of treatment
  The area under the curve (AUC) value determined by receiving operating characteristic (ROC) analysis of peripheral mitochondrial markers for the evolution of psychiatric symptoms following AD start, during a 8-weeks follow-up. Patients are identified as responders or nonresponders based on their clinical assessment
Predictive value for antidepressant response of MRI features | 8 weeks of treatment
  The area under the curve (AUC) value determined by receiving operating characteristic (ROC) analysis of MRI analysis for the evolution of psychiatric symptoms following AD start, during a 8-weeks follow-up. Patients are identified as responders or nonresponders based on their clinical assessment

IPD SHARING:
Plan to Share IPD: Undecided